CLINICAL TRIAL: NCT00323193
Title: Using MOVE! With Seriously Mentally Ill Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: D4219-R
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Mental Illness; Obesity
Keywords: Behavioral interventions; Mental Illness; Obesity; Psycho-educational interventions; Weight management
MeSH Terms: conditions — Mental Disorders; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): The intervention group completes approximately 8 individual level sessions with a MOVE specialist as well as approximately 8 group level intervention sessions.
  Interventions: Behavioral: MOVE!
- Arm 2 (No Intervention): The control group offers basic information about diet and exercise every month for six months.

INTERVENTIONS:
Behavioral: MOVE! — group based psychoeducation, motivation and support
  Arms: Arm 1

SUMMARY:
This study involves a controlled trial of an optimized version of a weight management and physical activity psycho-educational intervention (called MOVE!) with 200 obese and overweight veterans with serious mental illness.

DETAILED DESCRIPTION:
This study involves a controlled trial of an optimized version of a weight management and physical activity psycho-educational intervention (called MOVE!) for overweight and obese Veterans with serious mental illness. The study hypothesizes that MOVE! will result in weight loss and improved indicators of cardiovascular risk when compared to usual care. Medical outcomes are proportion achieving 4% or higher weight loss, mean weight loss, and reductions in cardiovascular risk (blood pressure, glucose and serum lipids). Psychosocial outcomes are general health, psychiatric functioning, quality of life, and self-esteem and medication adherence. Mediators include physical activity, dietary management, self-efficacy, and motivation/readiness to change. The intervention involves a well specified combination of individualized and group based services and draws on evidence based techniques and materials that are currently well packaged in an existing VA program called MOVE! The Comparison condition is operationalized as usual treatment plus monthly weight measurements and distribution of educational brochures regarding diet and exercise.

ELIGIBILITY:
Inclusion Criteria:

* DSM- IV diagnosis of schizophrenia spectrum disorders OR a DSM-IV diagnosis of other severe mental disorder including bipolar disorder, major depression, or severe anxiety disorder;
* Age between 18-64;
* No psychiatric hospitalization in 3-month period prior to enrollment;
* Community residency within 30 miles of either VA facility;
* A BMI of 25 or higher;
* Voluntary consent after receiving full information about the study;
* English speaking;
* Veteran of the armed forces

Exclusion Criteria:

* Active cancer other than non-melanoma skin cancer
* end stage chronic obstructive pulmonary disease
* end stage congestive heart failure
* end-stage neurological disorder
* problematic substance abuse as defined by provider
* end stage renal disease
* moderate to severe cognitive impairment (dementia, post-stroke)
* HIV positive with a CD4 count less than or equal to 350 within the last 6 months
* anorexia
* current pregnancy, currently nursing or planning to become pregnant in the next 6 months
* those living in long-term care facilities
* use in past 3 months of prescription pharmacological agents for weight loss
* no chart documented VA delivered medical primary care or general somatic care visit within the last 18 months
* most recent chart documented hematocrit level obtained within last six months is at or below 30%
* most recent chart documented creatinine level obtained within the last six months that is at or above 2.5
* most recent chart documented liver function tests obtained within the last six months exceeds twice the normal value for ALT, AST test in the Baltimore VA laboratory

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2006-07; Primary Completion 2010-01 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Goldberg, PhD, Principal Investigator — VA Maryland Health Care System, Baltimore
Locations (1):
- VA Maryland Health Care System, Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Result] Goldberg RW, Reeves G, Tapscott S, Medoff D, Dickerson F, Goldberg AP, Ryan AS, Fang LJ, Dixon LB. "MOVE!" Outcomes of a weight loss program modified for veterans with serious mental illness. Psychiatr Serv. 2013 Aug 1;64(8):737-44. doi: 10.1176/appi.ps.201200314. PMID 23584716

RESULTS

PARTICIPANT FLOW:
Groups:
- MOVE Group: The intervention group completes approximately 8 individual level sessions with a MOVE specialist as well as approximately 8 group level intervention sessions.
  MOVE!: group based psychoeducation, motivation and support
- Control Group: The control group offers basic information about diet and exercise every month for six months.
Period: Overall Study
Arm/Group | MOVE Group | Control Group
Started | 53 | 56
Completed | 30 | 41
Not Completed | 23 | 15

BASELINE CHARACTERISTICS:
Groups:
- Control Group: The control condition offers basic information about diet and exercise on a monthly basis.
- Total: Total of all reporting groups
Arm/Group | MOVE Group | Control Group | Total
Number analyzed (Participants) | 53 | 56 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 54 | 107
  >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 40 | 48 | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 36 | 29 | 65
  White | 16 | 21 | 37
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 53 | 56 | 109

OUTCOME MEASURES:

1. Primary Outcome: Weight Measurement
Description: Weight taken at the baseline assessment and again at the 6 month assessment
Time Frame: baseline and six months
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | MOVE Group | Control Group
Number analyzed (Participants) | 53 | 56
pounds
  Baseline Weight | 237.2 (50.3) | 230.2 (45.7)
  6 Month follow up | 240.8 (40.1) | 228.1 (43.4)
Statistical Analysis 1: Comparison: MOVE Group vs Control Group; Test type: Superiority or Other; p = .720, ANOVA

2. Secondary Outcome: Impact of Weight on Quality of Life Survey (IWQOL)
Description: Raw scores for this measure were converted to a range from 0 to 100, with higher scores indicating lower impact of weight on quality of life.
Time Frame: baseline and six months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MOVE Group | Control Group
Number analyzed (Participants) | 53 | 56
units on a scale
  Baseline | 67.6 (18.4) | 73.5 (21.4)
  6 Month Follow up | 75.1 (15.7) | 78.9 (19.1)
Statistical Analysis 1: Comparison: MOVE Group vs Control Group; Test type: Superiority or Other; p = .710, ANOVA

ADVERSE EVENTS:
Description: Adverse Events were reviewed for this study, although none were observed during the research trial.
Arm/Group | MOVE Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 0/53 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes